CLINICAL TRIAL: NCT03847896
Title: A 12-week, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group, Phase III Study Evaluating the Efficacy and Safety of PT027 Compared to PT008 and PT007 Administered QID in Adults and Children 4 Years of Age or Older With Asthma
Brief Title: A Study to Assess the Efficacy and Safety of Budesonide/Albuterol Metered Dose Inhaler (BDA MDI/PT027) Used 4 Times Daily in Adults and Children 4 Years of Age or Older With Asthma
Acronym: DENALI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV004; 2018-003674-27 (EudraCT Number)
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Results first posted 2022-09-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BDA MDI (PT027) 160/180 μg (Experimental): Budesonide/Albuterol sulfate BDA MDI (PT027) high dose
  Interventions: Combination Product: Budesonide/albuterol sulfate metered dose inhaler / BDA MDI 160/180 μg (high dose)
- BDA MDI (PT027) 80/180 μg (Experimental): Budesonide/Albuterol sulfate BDA MDI (PT027) low dose
  Interventions: Combination Product: Budesonide/albuterol sulfate metered dose inhaler / BDA MDI 80/180 μg (low dose)
- BD MDI (PT008) 160 µg (Active Comparator): Budesonide BD MDI (PT008)
  Interventions: Drug: Budesonide metered dose inhaler / BD MDI 160 µg
- AS MDI (PT007) 180 µg (Active Comparator): Albuterol sulfate AS MDI (PT007)
  Interventions: Drug: Albuterol sulfate metered dose inhaler / AS MDI 180 μg
- Placebo MDI (Placebo Comparator): Placebo MDI
  Interventions: Other: Placebo metered-dose inhaler / Placebo MDI

INTERVENTIONS:
Combination Product: Budesonide/albuterol sulfate metered dose inhaler / BDA MDI 160/180 μg (high dose) — Budesonide/albuterol sulfate pressurized metered dose inhaler (BDA MDI) 160/180 micrograms (μg), given as 2 inhalations of BDA MDI 80/90 μg, four times a day (QID)
  Arms: BDA MDI (PT027) 160/180 μg
Combination Product: Budesonide/albuterol sulfate metered dose inhaler / BDA MDI 80/180 μg (low dose) — Budesonide/albuterol sulfate pressurized metered dose inhaler (BDA MDI) 80/180 micrograms (μg), given as 2 inhalations of BDA MDI 40/90 μg, four times a day (QID)
  Arms: BDA MDI (PT027) 80/180 μg
Drug: Budesonide metered dose inhaler / BD MDI 160 µg — Budesonide pressurized metered dose inhaler (BD MDI) 160 micrograms (μg), given as 2 inhalations of BD MDI 80 μg, four times a day (QID)
  Arms: BD MDI (PT008) 160 µg
Drug: Albuterol sulfate metered dose inhaler / AS MDI 180 μg — Albuterol sulfate pressurized metered dose inhaler (AS MDI) 180 micrograms (μg), given as 2 inhalations of AS MDI 90 μg, four times a day (QID)
  Arms: AS MDI (PT007) 180 µg
Other: Placebo metered-dose inhaler / Placebo MDI — Placebo pressurized metered dose inhaler (Placebo MDI), given as 2 inhalations of Placebo MDI, four times a day (QID)
  Arms: Placebo MDI

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, parallel group study to compare 2 dose levels of budesonide/albuterol BDA MDI (PT027) to its components budesonide BD MDI (PT008) and albuterol AS MDI (PT007) on improvement in lung function and asthma symptoms after 12 weeks of treatment in adult, adolescent, and child subjects with symptomatic asthma currently being treated with a short/rapid-acting β2-adrenoreceptor agonist (SABA) as needed alone or with low-dose inhaled corticosteroid (ICS) maintenance therapy plus SABA as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged ≥4 years at the time of informed consent
2. Physician diagnosis of asthma with a documented history of the last 6 months
3. Receiving 1 of the following inhaled asthma medications with stable dosing for at least 30 days prior to Visit 1:

   * Only short/rapid-acting β2-adrenoreceptor agonist (SABA) used as needed
   * Stable low-dose inhaled corticosteroid in addition to as-needed use of SABA
4. Pre-bronchodilator FEV1 of ≥50 to <85% predicted normal value for adults (≥18 years of age) and ≥50% predicted normal value for subjects aged 4 to 17 years after withholding SABA ≥6 hours at Visit 1.
5. Demonstrate reversibility of airflow limitation defined as a ≥15% increase in FEV1 relative to baseline after administration of Sponsor-provided SABA (Ventolin) at either Visit 1 or Visit 1a.
6. Demonstrate acceptable spirometry performance acceptability/repeatability criteria
7. Taken Ventolin on ≥2 days out of 7 days prior to Visit 2
8. Demonstrate acceptable metered dose inhaler (MDI) administration technique as assessed by the investigator.
9. Able to perform acceptable and reproducible peak expiratory flow measurements as assessed by the investigator

Exclusion Criteria:

1. Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia)
2. Systemic corticosteroids (SCS) use (any dose and any indication) within 3 months before Visit 1
3. Chronic (≥3 weeks) use of SCS within 6 months prior to Visit 1
4. Received any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab) or investigational biologic within 3 months or 5 half-lives before Visit 1, whichever is longer, or any other prohibited medication
5. Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months before Visit 1 (including all forms of tobacco, e-cigarettes [vaping], and marijuana)
6. Life-threatening asthma defined as any history of significant asthma episode(s) requiring admission to an intensive care unit, intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s) within 5 years of Visit 1
7. Completed treatment for lower respiratory infection within 6 weeks prior to Visit 1
8. Upper respiratory infection involving antibiotic treatment not resolved within 7 days prior to Visit 1
9. Hospitalizations due to asthma within 6 months prior to Visit 1
10. Have taken ≥12 actuations per day of Sponsor-provided Ventolin during the run-in period prior to Visit 2 according to the below criteria:

    * ≥2 days out of 14 days of run-in
    * ≥3 days out of 15 to 21 days of run-in
    * ≥4 days out of 22 or more days of run-in
11. Unable to comply with study procedures including non-compliance with diary completion (ie, <70% subject completion of diary assessments in the last 7 days preceding Visit 2 or 4-times daily dosing, <80% compliance during the placebo run-in period).
12. Historical or current evidence of a clinically significant disease
13. Cancer not in complete remission for at least 5 years before Visit 1
14. Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 1
15. History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions if their magnitude is limiting informed consent validity
16. Significant abuse of alcohol or drugs, in the opinion of the investigator

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Albers, MD, PhD, Study Director — Avillion LLP
Locations (104):
- United States (63):
  - Research Site, Mobile, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Costa Mesa, California
  - Research Site, Encinitas, California
  - Research Site, Huntington Beach, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Greenacres City, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Woodbury, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Rolla, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Warrensburg, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Skillman, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Monroe, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Erie, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Gaffney, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Boerne, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Morgantown, West Virginia
  - Research Site, Greenfield, Wisconsin
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Czechia (7):
  - Research Site, Brandýs nad Labem
  - Research Site, Kralupy nad Vltavou
  - Research Site, Lovosice
  - Research Site, Neratovice
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Varnsdorf
- Germany (16):
  - Research Site, Berlin
  - Research Site, Darmstadt
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hessen
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Munich
  - Research Site, Neu-Isenburg
  - Research Site, Sachsen
  - Research Site, Schleswig
  - Research Site, Wiesbaden
  - Research Site, Witten
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Valjevo
- Slovakia (2):
  - Research Site, Košice
  - Research Site, Žilina
- Ukraine (9):
  - Research Site, Cherkasy
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chipps BE, Israel E, Beasley R, Panettieri RA Jr, Albers FC, Rees R, Dunsire L, Danilewicz A, Johnsson E, Cappelletti C, Papi A. Albuterol-Budesonide Pressurized Metered Dose Inhaler in Patients With Mild-to-Moderate Asthma: Results of the DENALI Double-Blind Randomized Controlled Trial. Chest. 2023 Sep;164(3):585-595. doi: 10.1016/j.chest.2023.03.035. Epub 2023 Mar 30. PMID 37003355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled on 20 March 2019 and the last subjected completed the study on 20 July 2021. Subjects were enrolled at 126 study centers worldwide (Argentina, Czechia, Germany, Serbia, Slovakia, Ukraine and the United States).
Pre-assignment Details: The randomized treatment phase started after a 2 to 4 week screening period during which participants self-administered single-blind Placebo MDI QID and Ventolin as needed to be used in response to asthma symptoms. In addition to the 1,001 subjects randomized, 875 subjects were screened but did not participate, of which 851 (97.3%) were ineligible, 3 were lost to follow up, 1 was excluded due to a protocol deviation, 18 withdrew by subject decision, and 2 withdrew by parent/guardian decision.
Period: Overall Study
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Started | 197 | 204 | 200 | 201 | 199
Completed | 190 | 188 | 188 | 184 | 178
Not Completed | 7 | 16 | 12 | 17 | 21
Not completed — Randomized in error and did not receive randomized study treatment | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 10 | 5 | 9 | 8
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 3 | 2 | 4
Not completed — A severe exacerbation event | 0 | 0 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Condition under investigation worsened | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 2
Not completed — Other reasons | 3 | 3 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 1,001 participants randomized, the full analysis set across all ages comprises 1,000 participants as one participant was randomized in error and did not receive study treatment. This participant has therefore been excluded from the summaries of baseline characteristics and efficacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI | Total
Number analyzed (Participants) | 197 | 204 | 199 | 201 | 199 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (15.80) | 48.7 (16.79) | 48.3 (15.80) | 47.0 (16.79) | 48.6 (15.82) | 48.5 (16.21)
Age, Customized [Count of Participants; unit: Participants]
  Children (>=4 to <12 years) | 0 | 3 | 0 | 4 | 3 | 10
  Adolescents (>=12 to <18 years) | 4 | 7 | 5 | 5 | 4 | 25
  Adults (>=18 to <65 years) | 154 | 155 | 161 | 159 | 161 | 790
  Elderly (>=65 years) | 39 | 39 | 33 | 33 | 31 | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 128 | 120 | 121 | 127 | 621
  Male | 72 | 76 | 79 | 80 | 72 | 379
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 62 | 50 | 46 | 63 | 282
  Not Hispanic or Latino | 136 | 142 | 149 | 155 | 136 | 718
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 1 | 3
  Asian | 1 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 15 | 18 | 30 | 19 | 96
  White | 179 | 185 | 180 | 167 | 174 | 885
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 1 | 3 | 4 | 14
Region of Enrollment [Number; unit: participants]
  Argentina | 9 | 11 | 14 | 14 | 6 | 54
  United States | 100 | 106 | 100 | 107 | 109 | 522
  Czechia | 12 | 12 | 12 | 17 | 18 | 71
  Ukraine | 44 | 44 | 43 | 32 | 40 | 203
  Slovakia | 1 | 0 | 0 | 0 | 0 | 1
  Serbia | 3 | 1 | 3 | 2 | 2 | 11
  Germany | 28 | 30 | 27 | 29 | 24 | 138
Height [Mean (Standard Deviation); unit: centimeters] | 167.8 (8.61) | 166.8 (9.71) | 167.7 (9.92) | 168.6 (9.86) | 168.0 (10.85) | 167.8 (9.81)
Weight [Mean (Standard Deviation); unit: kilograms] | 80.4 (16.43) | 80.0 (16.06) | 80.0 (14.52) | 82.3 (15.09) | 81.6 (17.79) | 80.9 (16.02)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.537 (5.2488) | 28.635 (4.8491) | 28.477 (4.9140) | 29.016 (4.8513) | 28.793 (5.2534) | 28.691 (5.0211)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Concentration Curve From 0 to 6 Hours (AUC0-6 Hours) Over 12 Weeks
Description: Lung function will be measured by spirometry. Baseline FEV1 will be taken as the average of the 60- and 30-minute pre-dose spirometry measures on or before randomization. Starting with the first study drug dose at Week 0 and then at Week 12, spirometry assessments will be completed at 60 and 30 minutes before the morning dose and 5, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes after dosing. FEV1 AUC0-6 hours will be calculated for changes from baseline (randomization visit) using the trapezoidal rule and will be normalized by dividing by the time (in hours) from dosing to the last measurement included (typically 6 hours).
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 197 | 200 | 199 | 195 | 196
milliliters | 258.6 (18.87) | 242.2 (18.80) | 178.0 (18.79) | 157.2 (19.08) | 96.7 (19.02)
Statistical Analysis 1: Comparison: AS MDI (PT007) 180 µg vs Placebo MDI; Only includes data from date of first dose up to date of last dose of randomized treatment. A sequential testing strategy is used such that the primary hypothesis tests are listed in ascending order of sequence. A null hypothesis can only be rejected if all preceding null hypotheses are also rejected. Tests are each conducted at the 5% level of significance; Test type: Superiority; p = 0.025, ANCOVA; Mean Difference (Final Values) = 60.5, 95% CI 2-sided [7.7 to 113.4]
Statistical Analysis 2: Comparison: BDA MDI (PT027) 160/180 μg vs Placebo MDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 161.9, 95% CI 2-sided [109.4 to 214.5]
Statistical Analysis 3: Comparison: BDA MDI (PT027) 160/180 μg vs BD MDI (PT008) 160 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = 80.7, 95% CI 2-sided [28.4 to 132.9]

2. Primary Outcome: Change From Baseline in Trough FEV1
Description: Trough FEV1 is calculated at each clinic visit as the average of the 30- and 60-minute pre-dose FEV1 measurements. Baseline FEV1 is defined as the average of the 30- and 60-minute pre-dose measures collected on the day of randomization.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 197 | 198 | 198 | 192 | 192
milliliters | 135.5 (24.58) | 123.5 (24.65) | 108.9 (24.51) | 2.7 (25.24) | 35.6 (25.12)
Statistical Analysis 1: Comparison: BD MDI (PT008) 160 µg vs Placebo MDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Final Values) = 73.3, 95% CI 2-sided [4.4 to 142.2]
Statistical Analysis 2: Comparison: BDA MDI (PT027) 160/180 μg vs Placebo MDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 99.9, 95% CI 2-sided [30.9 to 168.8]
Statistical Analysis 3: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 132.8, 95% CI 2-sided [63.6 to 201.9]
Statistical Analysis 4: Comparison: BDA MDI (PT027) 80/180 μg vs Placebo MDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.013, ANCOVA; Mean Difference (Final Values) = 87.9, 95% CI 2-sided [18.8 to 156.9]
Statistical Analysis 5: Comparison: BDA MDI (PT027) 80/180 μg vs AS MDI (PT007) 180 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 120.8, 95% CI 2-sided [51.5 to 190.1]

3. Secondary Outcome: Time to 15% Increase in FEV1 Over the Pre-treatment Value on Day 1
Description: The time to onset is defined as the time (minutes) from the first inhalation of randomized treatment (Day 1) to the first instance where a percentage change from baseline in FEV1 of at least 15% is observed. Participants were only to be included in the analysis if a percent change from baseline of at least 15% is observed within a nominal 30 minutes post dose assessment time point. Baseline FEV1 is defined as the average of the 30- and 60- minute pre-dose spirometry measures taken at randomization.
Time Frame: From first dose (first inhalation of randomized treatment) up to about 40 minutes post-dose (Day 1).
Population: Participants were only included in the analyses if a percent change from baseline of at least 15% is observed within the nominal 30 minutes post-dose.
Measure: Median (Full Range); unit: minutes
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 98 | 88 | 27 | 84 | 26
minutes | 7.5 [3 to 33] | 7.0 [3 to 35] | 17.0 [4 to 37] | 9.5 [4 to 37] | 14.0 [4 to 34]
Statistical Analysis 1: Comparison: AS MDI (PT007) 180 µg vs Placebo MDI; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -2.5, 95% CI 2-sided [-6 to 1]
Statistical Analysis 2: Comparison: BD MDI (PT008) 160 µg vs Placebo MDI; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = 3, 95% CI 2-sided [-3 to 9]
Statistical Analysis 3: Comparison: BDA MDI (PT027) 80/180 μg vs Placebo MDI; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -4.5, 95% CI 2-sided [-9 to 0]
Statistical Analysis 4: Comparison: BDA MDI (PT027) 160/180 μg vs Placebo MDI; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -4.5, 95% CI 2-sided [-9 to 0]
Statistical Analysis 5: Comparison: BDA MDI (PT027) 80/180 μg vs AS MDI (PT007) 180 µg; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -1.5, 95% CI 2-sided [-3 to 0]
Statistical Analysis 6: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -1, 95% CI 2-sided [-2 to 0]
Statistical Analysis 7: Comparison: BDA MDI (PT027) 80/180 μg vs BD MDI (PT008) 160 µg; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -6.5, 95% CI 2-sided [-11 to -2]
Statistical Analysis 8: Comparison: BDA MDI (PT027) 160/180 μg vs BD MDI (PT008) 160 µg; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = -6.5, 95% CI 2-sided [-11 to -2]
Statistical Analysis 9: Comparison: BDA MDI (PT027) 160/180 μg vs BDA MDI (PT027) 80/180 μg; Not type-I error controlled. The estimated median difference and 95% CIs are calculated using the Hodges-Lehmann method; Test type: Superiority; Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1]

4. Secondary Outcome: Duration of 15% Increase in FEV1 Over the Pre-treatment Value on Day 1
Description: The duration of onset is defined as the time (minutes) of the continual period in which a percentage increase change from baseline in FEV1 of at least 15% is observed. Participants will only be included in the analyses if a percent change from baseline of at least 15% is observed within a nominal 30 minutes post dose assessment. If a participant has multiple periods of onset, only the first will contribute to the summary. Duration of onset can last up to the last assessment during a nominal 6 hour serial spirometry profile. Baseline FEV1 is defined as the average of the 60- and 30- minute pre-dose spirometry taken at randomization.
Time Frame: Onset up to about 40 minutes post-treatment, with duration lasting up to the last assessment of a nominal 6 hour serial spirometry profile (Day 1).
Measure: Median (Full Range); unit: Minutes
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 98 | 88 | 27 | 84 | 26
Minutes | 185.5 [4 to 363] | 174 [10 to 362] | 98 [14 to 354] | 158.5 [9 to 363] | 229.5 [8 to 356]

5. Secondary Outcome: Number of Participants With a Clinically Meaningful Difference on the Asthma Control Questionnaire 7-item Version (ACQ-7) at Week 12.
Description: A responder is defined as a participant who achieves a reduction from baseline in overall ACQ-7 score of at least 0.5. The ACQ-7 has 7 questions, with each question using a 7 point scale, where 0 = totally controlled and 6 = extremely poorly controlled. The overall ACQ-7 score is defined as the averaged score across the 7 questions. The analysis only includes participants who are uncontrolled at basellne, i.e. baseline ACQ-7 >= 1.5. All participants who discontinue treatment prior to Week 12 are classified as non-responders.
Time Frame: Baseline and 12 weeks
Population: The analysis only includes participants who are uncontrolled at baseline, i.e. ACQ-7 >= 1.5. All participants who discontinue treatment prior to Week 12 are classified as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 161 | 165 | 162 | 163 | 159
Participants | 107 | 108 | 100 | 77 | 88
Statistical Analysis 1: Comparison: AS MDI (PT007) 180 µg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.118, Regression, Logistic; Odds Ratio (OR) = 0.699, 95% CI 2-sided [0.445 to 1.096]
Statistical Analysis 2: Comparison: BD MDI (PT008) 160 µg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.161, Regression, Logistic; Odds Ratio (OR) = 1.386, 95% CI 2-sided [0.878 to 2.187]
Statistical Analysis 3: Comparison: BDA MDI (PT027) 80/180 μg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.044, Regression, Logistic; Odds Ratio (OR) = 1.605, 95% CI 2-sided [1.013 to 2.541]
Statistical Analysis 4: Comparison: BDA MDI (PT027) 160/180 μg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.039, Regression, Logistic; Odds Ratio (OR) = 1.626, 95% CI 2-sided [1.024 to 2.584]
Statistical Analysis 5: Comparison: BDA MDI (PT027) 80/180 μg vs AS MDI (PT007) 180 µg; Comparison is not type-I error controlled; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.297, 95% CI 2-sided [1.456 to 3.626]
Statistical Analysis 6: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Comparison is not type-I error controlled; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.328, 95% CI 2-sided [1.471 to 3.687]
Statistical Analysis 7: Comparison: BDA MDI (PT027) 80/180 μg vs BD MDI (PT008) 160 µg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.532, Regression, Logistic; Odds Ratio (OR) = 1.158, 95% CI 2-sided [0.731 to 1.835]
Statistical Analysis 8: Comparison: BDA MDI (PT027) 160/180 μg vs BD MDI (PT008) 160 µg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.499, Regression, Logistic; Odds Ratio (OR) = 1.174, 95% CI 2-sided [0.737 to 1.868]
Statistical Analysis 9: Comparison: BDA MDI (PT027) 160/180 μg vs BDA MDI (PT027) 80/180 μg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.955, Regression, Logistic; Odds Ratio (OR) = 1.014, 95% CI 2-sided [0.635 to 1.618]

6. Secondary Outcome: Change From Baseline in Trough FEV1 at Week 1.
Description: Trough FEV1 is calculated at each clinic visit as the average of the 60- and 30-minute pre-dose FEV1 measurements. Baseline FEV1 is defined as the average of the 60- and 30-minute pre-dose measures collected on the day of randomization.
Time Frame: Baseline and 1 week
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
Number analyzed (Participants) | 197 | 198 | 198 | 192 | 192
milliliters | 107.2 (21.46) | 72.0 (21.31) | 93.4 (21.35) | -0.8 (21.69) | 41.3 (21.47)
Statistical Analysis 1: Comparison: AS MDI (PT007) 180 µg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.169, ANCOVA; Mean Difference (Final Values) = -42.1, 95% CI 2-sided [-101.9 to 17.8]
Statistical Analysis 2: Comparison: BD MDI (PT008) 160 µg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.086, ANCOVA; Mean Difference (Final Values) = 52.1, 95% CI 2-sided [-7.4 to 111.5]
Statistical Analysis 3: Comparison: BDA MDI (PT027) 80/180 μg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.31, ANCOVA; Mean Difference (Final Values) = 30.7, 95% CI 2-sided [-28.6 to 90.1]
Statistical Analysis 4: Comparison: BDA MDI (PT027) 160/180 μg vs Placebo MDI; Comparison is not type-I error controlled; Test type: Superiority; p = 0.03, ANCOVA; Mean Difference (Final Values) = 65.9, 95% CI 2-sided [6.3 to 125.4]
Statistical Analysis 5: Comparison: BDA MDI (PT027) 80/180 μg vs AS MDI (PT007) 180 µg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.017, ANCOVA; Mean Difference (Final Values) = 72.8, 95% CI 2-sided [13.1 to 132.5]
Statistical Analysis 6: Comparison: BDA MDI (PT027) 160/180 μg vs AS MDI (PT007) 180 µg; Comparison is not type-I error controlled; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 107.9, 95% CI 2-sided [48.1 to 167.8]
Statistical Analysis 7: Comparison: BDA MDI (PT027) 80/180 μg vs BD MDI (PT008) 160 µg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.48, ANCOVA; Mean Difference (Final Values) = -21.3, 95% CI 2-sided [-80.5 to 37.9]
Statistical Analysis 8: Comparison: BDA MDI (PT027) 160/180 μg vs BD MDI (PT008) 160 µg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.648, ANCOVA; Mean Difference (Final Values) = 13.8, 95% CI 2-sided [-45.6 to 73.2]
Statistical Analysis 9: Comparison: BDA MDI (PT027) 160/180 μg vs BDA MDI (PT027) 80/180 μg; Comparison is not type-I error controlled; Test type: Superiority; p = 0.246, ANCOVA; Mean Difference (Final Values) = 35.1, 95% CI 2-sided [-24.2 to 94.5]

ADVERSE EVENTS:
Time Frame: Approximately 12 weeks.
Description: Adverse events were collected from the time of signed informed consent/assent and up to the safety follow up period. Reported adverse events are those that occurred from the date of first dose of randomized treatment up to the date of treatment discontinuation.
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | BD MDI (PT008) 160 µg | AS MDI (PT007) 180 µg | Placebo MDI
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/204 | 0/199 | 0/201 | 0/199
Serious Adverse Events (participants affected / at risk) | 2/197 | 4/204 | 3/199 | 1/201 | 3/199
Other Adverse Events (participants affected / at risk) | 37/197 | 31/204 | 31/199 | 29/201 | 38/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=197) | BDA MDI (PT027) 80/180 μg (N=204) | BD MDI (PT008) 160 µg (N=199) | AS MDI (PT007) 180 µg (N=201) | Placebo MDI (N=199)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=197) | BDA MDI (PT027) 80/180 μg (N=204) | BD MDI (PT008) 160 µg (N=199) | AS MDI (PT007) 180 µg (N=201) | Placebo MDI (N=199)
Nasopharyngitis (Infections and infestations) | 15 | 13 | 10 | 9 | 11
Headache (Nervous system disorders) | 10 | 10 | 7 | 11 | 14
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 5 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 2 | 0
Hypertension (Vascular disorders) | 4 | 2 | 0 | 2 | 2
COVID-19 (Infections and infestations) | 2 | 1 | 1 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data or results obtained from this study must not be published without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03847896/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03847896/SAP_001.pdf